CLINICAL TRIAL: NCT05067543
Title: Perform Humeral System Study
Acronym: PHS
Status: Recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 20D-W-PHS-RM
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis Shoulder; Avascular Necrosis; Post-traumatic Arthrosis of Other Joints, Shoulder Region; Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Osteonecrosis; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Tornier Perform Humeral System - Stem: Partial or total shoulder arthroplasty using the Tornier Perform Humeral Stem.
  Interventions: Device: Tornier Perform Humeral - Stem

INTERVENTIONS:
Device: Tornier Perform Humeral - Stem — The PERFORM Humeral System - Stem is a non-constrained prosthesis intended for the total or partial replacement of the glenohumeral articulation.

SUMMARY:
This study is an international, single arm, multicenter, prospective, non-significant risk, Post-Market Clinical Follow-up study, which is designed to collect safety and performance data at baseline, surgery, immediate post-op and annually through 10 years post-operation.

Data collected from this study will be used for purposes, including but not limited to, Post-Market Surveillance, peer-reviewed publications, education materials, regulatory submissions, and/or product development.

DETAILED DESCRIPTION:
This study is an international, single arm, multicenter, prospective, non-significant risk, Post-Market Clinical Follow-up study. Data will be collected for the commercially available PERFORM™ Humeral System. The objective of this study is to demonstrate the safety and performance of the PERFORM™ Humeral System devices after implantation over a standard follow-up period using Patient Reported Outcome Measures related to quality of life, pain and functional improvements, safety of the implants, as well as radiographic assessments. Safety and performance measures will be evaluated throughout the patient's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of the informed consent or non-opposition (when applicable).
* Informed and willing to sign an informed consent form approved by IRB or EC (when applicable).
* Willing and able to comply with the requirements of the study protocol.
* Considered a candidate for shoulder arthroplasty using a study device.
* Meets indications for use requirements or other local, regional, or geographic specific regulatory requirements

Exclusion Criteria:

* Not able to comply with the study procedures based on the judgment of the assessor (e.g. cannot comprehend study questions, inability to keep scheduled assessment times)
* Patient belongs to a vulnerable group of patients, including minor patients, those unable to decide for themselves to participate or needing a Legally Authorized Representative (LAR), or others who could be subject to coercion (patients who may not be acting on their own initiative) (referred as "vulnerable subject" in the section 3.44 of the ISO 14155 norm).
* Active local or systemic infection, sepsis, or osteomyelitis
* Poor bone quality, where there could be considerable migration of the prothesis and/or a chance of fracture of the humerus or glenoid
* Significant injury to the brachial plexus
* Inadequate bone stock in the proximal humerus or glenoid fossa for supporting the components
* Neuromuscular disease (e.g., joint neuropathy)
* Patient with known allergy to one of the product materials
* Metabolic disorders which may impair bone formation
* Patient pregnancy
* Planned for two-stage surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients intended for the total or partial replacement of the glenohumeral articulation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2035-06-30 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to last follow-up visit in ASES scores | Baseline through Follow-Up visits through 24 months Post-Op
  ASES Score = American Shoulder and Elbow Surgeons Score, 11 items with total score reported out of 100 measuring pain and activity of patient's evaluated shoulder where lower scores indicate more pain and less function

SECONDARY OUTCOMES:
Change from Baseline to last follow-up visit in Constant Murley scores | Baseline through Follow-Up visits through 10 years Post-Op
  Combination of physician-completed and patient-reported portions to assess functional state of shoulder including range of motion; total score reported out of 100 measuring where lower scores indicate less function of the evaluated shoulder
Change from Baseline to last follow-up visit in SANE scores | Baseline through Follow-Up visits through 10 years Post-Op
  SANE = Single Assessment Numeric Evaluation; 1 item assessment of shoulder rating 0% to 100%
Change from Baseline to last follow-up visit in Subject Satisfaction scores | Baseline through Follow-Up visits through 10 years Post-Op
  Single, subjective question measuring patient satisfaction; assessed by improved, worsened, or no change in satisfaction
Change from Baseline to last follow-up visit in EQ-5D scores | Baseline through Follow-Up visits through 10 years Post-Op
  The EuroQol Five Dimensions Questionnaire (EQ-5D) questionnaire is a standardized instrument for use as a measure of quality of life. It is cognitively simple, takes only a few minutes to complete, and provides a simple descriptive profile as well as a single index value for quality of life that can be used in the clinical and economic evaluation of health care. The EQ-5D consists of a descriptive system which comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression), and a visual analog scale which measures the respondent's self-rated health on a 0-100 scale.
Number of device associated and procedure associated adverse events. | Baseline through Follow-Up visits through 10 years Post-Op
Rates of revision surgeries. | Baseline through Follow-Up visits through 10 years Post-Op
Evaluation of radiological imaging of the affected shoulder | Baseline through Follow-Up visits through 10 years Post-Op
  Images will be analyzed for bone characteristics (baseline and post-op) and device migration, component breakage, and radiolucency (post-op visits only).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma
Locations (10):
- United States (6):
  - Baptist Healthcare, Lexington, Kentucky
  - Summit Orthopedics, Eagan, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Orthopedic Institute, Sioux Falls, South Dakota
  - University of Utah, Salt Lake City, Utah
- Roth McFarlane Hand and Upper Limb Centre, London, Ontario, Canada
- Orthopedic Center Santy, Lyon, France
- Schulthess Klinik, Zurich, Switzerland
- Wrightington Hospital, Wigan, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No